CLINICAL TRIAL: NCT00744484
Title: A 12 Week Physical Training Programme for Patients With Chronic Obstructive Pulmonary Disease (COPD)-a Comparison of Water Based and Land Based Group Training
Brief Title: A 12 Week Physical Training Programme for Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other); Nord-Trøndelag University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4.2007.679 (REK); 17117 (Other: NSD)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Physical group training; Water exercise; Cardiorespiratory fitness; Functional exercise capacity; Health related quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B1 (Experimental): B1 - training in water
  Interventions: Behavioral: Training in water
- S1 (Experimental): S1 - training on land
  Interventions: Behavioral: Training on land

INTERVENTIONS:
Behavioral: Training in water — 45 minutes interval training in water, submaximal intensity, twice a week
  Arms: B1
Behavioral: Training on land — 45 minutes interval training on land, submaximal intensity, twice a week
  Arms: S1

SUMMARY:
The purpose of this study is to determine whether water based or land based group training is more effective for people with COPD.

DETAILED DESCRIPTION:
COPD is a more common diagnosis today compared to 20 years ago, and the group is growing fast. The suffering caused by COPD and the financial cost to society is on the increasing. The principal causes of COPD are smoking and inactivity. So far it is poorly understood wich form of exercise is the most effective in training this condition.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD II
* Not taking part in physical activity during the last year

Exclusion Criteria:

* COPD GOLD I, III, IV
* Pain in the legs that make activity difficult

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
VO2 peak | 12 weeks

SECONDARY OUTCOMES:
Health related quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thor Naustdal, MD, Principal Investigator — Hospital of Levanger / NTNU ISB
Locations (1):
- Levanger Hosp, Levanger, Nord-Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: No